CLINICAL TRIAL: NCT01354717
Title: Phase 3 Study of Brand Generic and Placebo in Treatment of Actinic Keratosis
Brief Title: Bioequivalence Study of Generic Fluorouracil 0.5% Cream and 0.5% Carac® and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spear Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Spear 0.5%
Record Dates: First submitted 2011-05-14; First posted 2011-05-17 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil; Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brand Carac (Active Comparator): Treatment of actinic keratosis with active ingredient
  Interventions: Drug: Brand Carac
- Generic 0.5% 5-fluorouracil cream (Active Comparator): Treatment of actinic keratosis with active ingredient
  Interventions: Drug: Generic 0.5% 5-fluorouracil cream
- Placebo (Placebo Comparator): treatment of actinic keratosis with placebo cream
  Interventions: Other: Placebo cream

INTERVENTIONS:
Drug: Brand Carac — treatment of actinic keratosis
  Other Names: 5-fu
  Arms: Brand Carac
Drug: Generic 0.5% 5-fluorouracil cream — treatment of actinic keratosis
  Other Names: 5-fu
  Arms: Generic 0.5% 5-fluorouracil cream
Other: Placebo cream — treatment of actinic keratosis
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, three treatment parallel study in which normal, healthy men and women (age 45-85) with actinic keratosis will be treated on the face once daily for two weeks with 5-Fluorouracil Cream 0.5%, Spear Pharmaceuticals (Generic), Carac® Cream 0.5% (Brand), or Cream Vehicle (Placebo). Actinic keratoses will be counted at the baseline visit and at the visit four weeks following cessation of treatment.

DETAILED DESCRIPTION:
actinic keratosis

ELIGIBILITY:
Inclusion Criteria:

Men and women with the presence of actinic keratoses

* Women who have had surgical sterilization or are post-menopausal (absence of menses for at least one year) are eligible. Women of child-bearing potential who are non-pregnant and non-nursing, and willing to avoid pregnancy during the course of the study and during the menstrual cycle following completion of their participation in the study are eligible. (Adequate contraception is defined as regular use of, diaphragm with condoms, IUD with condoms, or systemic contraceptives - if used for at least three months prior to enrollment in the study). A negative pregnancy test is required at entry into the study
* Able to refrain from the use of all other topical medications to the facial area during the treatment period
* Considered reliable and capable of understanding their responsibility and role in the study
* Have provided written informed consent

Exclusion Criteria:

* History of allergy or hypersensitivity to 5-fluorouracil

  * Known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency
  * Clinical evidence of severe, uncontrolled auto-immune, cardiovascular, gastrointestinal, hematological, hepatic, neurological, pancreatic, pulmonary or renal disease
  * Dermatologic conditions if present on the face such as: atopic dermatitis, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, or albinism
  * Positive urine pregnancy test in women of child-bearing potential
  * Inability to use adequate birth control measures for women of child-bearing potential, as defined above
  * Serious psychological illness
  * Significant history (within the past year) of alcohol or drug abuse
  * Participation in any clinical research study during the 30 day period preceding study initiation
  * Medical history which, based on the clinical judgment of the investigator, implies an unlikelihood of successful completion of the study
  * Treatment for actinic keratosis or skin cancer in the previous 28 days with the following: topical 5 fluorouracil, cryodestruction (liquid nitrogen spray), curettage (scraping of pre-cancer or skin cancers), surgical removal of skin cancer, photodynamic therapy, surgical excision, topical diclofenac (Solaraze), topical imiquimod (Aldara), topical retinoids if used for actinic keratosis or other treatments for actinic keratoses
  * Application of 1) chemical peel, 2) dermabrasion, 3) laser abrasion, 4) PUVA (psoralen plus ultraviolet A) therapy, or 5) UVB therapy to the face or bald scalp within six months prior to randomization
  * Use of sun lamps or sun tanning beds or booths during the 2 weeks prior to first application until Day 42 visit
  * Any oral (systemic steroids) or topical corticosteroids within 1 month of study entry, except for subjects on chronic low dose corticosteroids less than 5 mg daily for greater than 1 year
  * Use within 1 month of any immunomodulators like interferon, or cytotoxic drugs
  * Prior treatment with systemic 5-fluorouracil or systemic cancer therapy within 6 months of study entry
  * Subjects with lesions suspicious for squamous cell carcinoma

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Percent of patients with clearing | August 28, 2010 to March 17, 2011
Clearing of actinic keratosis | 42 days

SECONDARY OUTCOMES:
superiority to placebo | 42 days

OTHER OUTCOMES:
Irritation | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Appell, M.D., Principal Investigator — Alliance Clinical Research, Inc